CLINICAL TRIAL: NCT05422716
Title: "Epidural Spinal Cord Stimulation: Addressing Spasticity and Motor Function"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-1176-22
Record Dates: First submitted 2022-05-05; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Spasticity
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: participants will be randomized into either the baclofen group or epidural stimulation
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgically implanted epidural stimulation for spasticity (Experimental): The epidural stimulation (ES) group will undergo the research protocol for epidural stimulator surgical implant followed by mapping studies to identify targeted stimulation configurations for spasticity. In each subsequent 6 months we will enroll cohorts of (n=5) voluntary research participants to allow for the final cohort to complete their 6 month follow up with a remaining 3 months for final data analyses and dissemination for the grant period.
  Spinal cord epidural stimulation is administered by a multi-electrode array implanted in the epidural space over the dorsum of the spinal cord.
  Interventions: Device: Epidural implant stimulation device
- Surgically implanted Intrathecal baclofen pump, the standard of care control group (Experimental): Individuals randomized to the baclofen pump (BP) group will continue with their clinical surgical and maintenance plan while also participating in all of the outcomes (assessments).
  The Baclofen pump will be surgically implanted by a member of the clinical SCI medical team.
  Interventions: Device: Epidural implant stimulation device

INTERVENTIONS:
Device: Epidural implant stimulation device — Individuals randomized to the Baclofen pump device group will continue with their clinical surgical and maintenance plan while also participating in all of the outcomes (assessments). The epidural implant group will undergo the research protocol for epidural stimulator surgical implant followed by mapping studies to identify targeted stimulation configurations for spasticity.
  Other Names: Baclofen Pump device

SUMMARY:
This study aims to expand the knowledge and capacity for neuromodulation to improve the debilitating effects of severe spasticity (spasms, tonic muscle activity and/or clonus) in persons with spinal cord injury (SCI). The purpose of this study is to compare if spinal cord epidural stimulation can treat severe spasticity more effectively and have fewer side effects than a baclofen pump.

DETAILED DESCRIPTION:
This study aims to expand our knowledge and capacity for neuromodulation to improve the debilitating effects of severe spasticity (spasms, tonic muscle activity and/or clonus) in persons with spinal cord injury (SCI) who are not adequately treated with oral pharmacological management, while avoiding side effects, and also improving voluntary control using surgically implantable targeted tonic spinal cord epidural stimulation (scES) . Individuals recruited and enrolled in the study will have significant spasticity not adequately treated by oral medications and clinically referred for an intrathecal baclofen pump trial. Current treatment of severe spasticity by pharmacological treatments are associated with several concomitant side effects that have consequences including limiting the ability to participate in and respond to neurorehabilitation15 and diminishing quality of life. Also, for persons with SCI and severe spasticity, available rehabilitation therapies are limited in their ability to foster appropriate neural excitation and subsequently motor recovery.

This study focuses on ameliorating severe spasticity through specific spasticity-targeted spinal cord epidural stimulation (SP-scES) that has been shown to mediate levels of neural excitation for movement and unwanted muscle activation. The study will be evaluated as compared to a standard of care control group using pharmacological administration via an intrathecal baclofen pump (ITBP). In the long-term, this study will also provide a framework to develop clinically viable approaches with tools to provide optimized care for individuals with chronic SCI. This research is directly aimed to improve the quality of life for those affected by and living with SCI by reducing spasticity (and increasing voluntary control of movement) in the home and community while avoiding debilitating side effects of long-term pharmacological intervention.

ELIGIBILITY:
Inclusion Criteria:

1. I must be at least 18 years of age
2. I must have a non-progressive spinal cord injury (SCI)
3. I have met the clinical criteria for an intrathecal baclofen pump
4. I am in stable medical condition

Exclusion Criteria:

1. I must not be ventilator dependent
2. I must not have untreated painful musculoskeletal dysfunction, fracture or pressure injury
3. I must not have untreated psychiatric disorder or ongoing drug abuse, as determined by study staff
4. I must not have cardiac, respiratory, bladder, renal or other untreated medical disorder unrelated to SCI
5. I must not have had peripheral muscle Botox injections less than 12 months prior to implant
6. I must not have a colostomy bag or urostomy
7. I must not have any implanted pump (i.e., baclofen pump, pain pump, etc.) prior to randomization
8. I must not be pregnant at the time of enrollment or planning to become pregnant during the time course of the study
9. I must not have an active implantable device that may interfere with the epidural neurostimulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-14 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Quantification of muscle Activity Using Integrated EMG in Response to Triggered Spasticity | Baseline assessment through study completion, an average of 8 months. Assessments will be preformed: prior to being implanted and 3 months and 6 months after implantation)
  Three common triggers of spasticity for each person will be identified, such as quick stretch of the ankle, flexion/extension of the hip, and rapid position changes. Each trigger will be implemented consecutively three times while recording EMG from the hip, knee, and ankle muscles bilaterally. Integrated EMG will assess the total EMG activity generated in response to the spasticity trigger for each muscle for each attempt. Muscles: (SOL), medial gastrocnemius (MG), tibialis anterior (TA), medial hamstrings (MH), quadriceps (VL and RF), adductor (AD) and/or other related muscles.

SECONDARY OUTCOMES:
The Penn Spasm Scale | Baseline assessment through study completion, an average of 8 months. Assessments will be preformed: prior to being implanted and 3 months and 6 months after implantation)
  The Penn Spasm Scale is a self-report noting both the severity and frequency of spasms
Modified Ashworth Score | Baseline assessment through study completion, an average of 8 months. Assessments will be preformed: prior to being implanted and 3 months and 6 months after implantation)
  Modified Ashworth Score assesses on a scale of 0 to 4 the resistance of a relaxed, single joint as it is moved throughout its full available range of motion. Participants will be instructed to relax and to allow the examiner to perform the test movements
Frequency of Side Effects | Baseline assessment through study completion, an average of 8 months. Assessments will be preformed: prior to being implanted and 3 months and 6 months after implantation)
  The side effects including fatigue, drowsiness, dizziness, weakness, confusion, headache, nausea, and sexual dysfunction will be recorded using temporaneous recording of each effect and its duration with STIMX PICS algorithms.
  STIMX PICS recordings (subjective spasticity measures and frequency of side effects) will occur for 24 hours twice prior to implantation and weekly after surgery throughout the 3 months of intervention.
Quantification of Muscle Activity Using Integrated EMG in Response to Voluntary Leg Movement | Baseline assessment through study completion, an average of 8 months. Assessments will be preformed: prior to being implanted and 3 months and 6 months after implantation)
  Hip and knee extension and flexion and ankle dorsi and plantar flexion will be attempted consecutively three times in response to a 3 tone while recording EMG from the hip, knee, and ankle muscles bilaterally.
NeuroRecovery Scale (NRS) for Lower Body and Trunk | Baseline assessment through study completion, an average of 8 months. Assessments will be preformed: prior to being implanted and 3 months and 6 months after implantation)
  The NRS is a valid, reliable, and responsive evaluation tool for measuring functional recovery in persons with SCI based on tasks that test pre-injury functional capability.
The AIS Impairment Scale | Baseline assessment through study completion, an average of 8 months. Assessments will be preformed: prior to being implanted and 3 months and 6 months after implantation)
  The ASIA Impairment Scale (AIS) is a classification in SCI that describes the level and severity of the injury, based upon the motor and sensory examination as described in the International Standards of Neurological Classification for SCI (ISNCSCI)

IPD SHARING:
Plan to Share IPD: No